CLINICAL TRIAL: NCT02787213
Title: A Multicenter Assessment of a Spontaneous Preterm Birth Risk Predictor
Acronym: TREETOP
Status: Completed | Type: Observational
Sponsor: Sera Prognostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SP 014
Record Dates: First submitted 2016-05-17; First posted 2016-06-01 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Preterm Birth
Keywords: proteomics; pregnancy; biomarkers; preterm birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Women with preterm delivery
- Women without preterm delivery

SUMMARY:
Prospective multicenter observational study to further develop and validate a preterm birth risk predictor, using a preterm cutoff at 37 0/7 weeks gestation and at 35 0/7 weeks gestation. A single maternal peripheral blood sample will be collected for analysis. Data related to potential risk factors for preterm birth will be obtained through maternal interview and review of medical records. Subjects will be followed through the delivery process to assess the course of pregnancy, labor, and to document any related maternal complications. Neonatal outcomes will be gathered from the medical record for up to 28 days of life or discharge, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject has singleton gestation
* Subject is able to provide consent
* Gestational age is confirmed by a documented crown rump length on an ultrasound performed at the study site within 6 0/7 weeks and 13 6/7 weeks gestation (first trimester)
* Subject has no signs and/or symptoms of preterm labor and has intact membranes
* Investigator believes subject is willing to comply with study visits and procedures
* Investigator believes the subject's delivery data will be available within 15 business days from delivery, and neonatal data will be available for data collection purposes within 15 business days from discharge

Exclusion Criteria:

* The subject has a planned cesarean section or induction of labor prior to 370/7 weeks of gestation
* The subject has a planned cerclage placement for the current pregnancy
* There is a known or suspected fetal anomaly or chromosomal abnormality
* The subject has had a blood transfusion during the current pregnancy
* The subject has known elevated bilirubin levels (hyperbilirubinemia)
* The subject has taken or plans to take any of the following medications during the current pregnancy:

  * Progesterone or progesterone-derivative medication after 13 6/7 weeks gestation
  * Enoxaparin, heparin, heparin sodium, low molecular weight heparin after first day of last menstrual period
* The subject has participated in, or plans to participate in, an interventional treatment study during the current pregnancy
* The current pregnancy was previously a multiple gestation that is now a single fetus due to reduction, vanishing twin, etc.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women, 18 years or older, who are receiving prenatal care.
Sampling Method: Probability Sample
Enrollment: 5011 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operator characteristic curve (AUROC) for prediction of preterm versus term birth using freshly collected specimens. | Up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Durlin E Hickok, MD, Study Chair — Sera Prognostics
Locations (18):
- United States (18):
  - Maricopa Integrated Health Systems, Phoenix, Arizona
  - University of California, Irvine Medical Center, Orange, California
  - UC San Diego Health, San Diego, California
  - University of Colorado-Denver, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Sciences University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Regional Obstetrical Consultants, Chattanooga, Tennessee
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared once it is published.

REFERENCES:
- [Background] Saade GR, Boggess KA, Sullivan SA, Markenson GR, Iams JD, Coonrod DV, Pereira LM, Esplin MS, Cousins LM, Lam GK, Hoffman MK, Severinsen RD, Pugmire T, Flick JS, Fox AC, Lueth AJ, Rust SR, Mazzola E, Hsu C, Dufford MT, Bradford CL, Ichetovkin IE, Fleischer TC, Polpitiya AD, Critchfield GC, Kearney PE, Boniface JJ, Hickok DE. Development and validation of a spontaneous preterm delivery predictor in asymptomatic women. Am J Obstet Gynecol. 2016 May;214(5):633.e1-633.e24. doi: 10.1016/j.ajog.2016.02.001. Epub 2016 Feb 11. PMID 26874297
- [Background] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Background] Goldenberg RL, Rouse DJ. Prevention of premature birth. N Engl J Med. 1998 Jul 30;339(5):313-20. doi: 10.1056/NEJM199807303390506. No abstract available. PMID 9682045
- [Background] Rush RW, Keirse MJ, Howat P, Baum JD, Anderson AB, Turnbull AC. Contribution of preterm delivery to perinatal mortality. Br Med J. 1976 Oct 23;2(6042):965-8. doi: 10.1136/bmj.2.6042.965. PMID 974709
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Gravett MG, Novy MJ, Rosenfeld RG, Reddy AP, Jacob T, Turner M, McCormack A, Lapidus JA, Hitti J, Eschenbach DA, Roberts CT Jr, Nagalla SR. Diagnosis of intra-amniotic infection by proteomic profiling and identification of novel biomarkers. JAMA. 2004 Jul 28;292(4):462-9. doi: 10.1001/jama.292.4.462. PMID 15280344
- [Background] Ruetschi U, Rosen A, Karlsson G, Zetterberg H, Rymo L, Hagberg H, Jacobsson B. Proteomic analysis using protein chips to detect biomarkers in cervical and amniotic fluid in women with intra-amniotic inflammation. J Proteome Res. 2005 Nov-Dec;4(6):2236-42. doi: 10.1021/pr050139e. PMID 16335971
- [Background] Buhimschi CS, Bhandari V, Hamar BD, Bahtiyar MO, Zhao G, Sfakianaki AK, Pettker CM, Magloire L, Funai E, Norwitz ER, Paidas M, Copel JA, Weiner CP, Lockwood CJ, Buhimschi IA. Proteomic profiling of the amniotic fluid to detect inflammation, infection, and neonatal sepsis. PLoS Med. 2007 Jan;4(1):e18. doi: 10.1371/journal.pmed.0040018. PMID 17227133
- [Background] Gravett MG, Thomas A, Schneider KA, Reddy AP, Dasari S, Jacob T, Lu X, Rodland M, Pereira L, Sadowsky DW, Roberts CT Jr, Novy MJ, Nagalla SR. Proteomic analysis of cervical-vaginal fluid: identification of novel biomarkers for detection of intra-amniotic infection. J Proteome Res. 2007 Jan;6(1):89-96. doi: 10.1021/pr060149v. PMID 17203952
- [Background] Pereira L, Reddy AP, Jacob T, Thomas A, Schneider KA, Dasari S, Lapidus JA, Lu X, Rodland M, Roberts CT Jr, Gravett MG, Nagalla SR. Identification of novel protein biomarkers of preterm birth in human cervical-vaginal fluid. J Proteome Res. 2007 Apr;6(4):1269-76. doi: 10.1021/pr0605421. Epub 2007 Mar 21. PMID 17373840
- [Background] Esplin MS, Merrell K, Goldenberg R, Lai Y, Iams JD, Mercer B, Spong CY, Miodovnik M, Simhan HN, van Dorsten P, Dombrowski M; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Proteomic identification of serum peptides predicting subsequent spontaneous preterm birth. Am J Obstet Gynecol. 2011 May;204(5):391.e1-8. doi: 10.1016/j.ajog.2010.09.021. Epub 2010 Nov 11. PMID 21074133
- [Background] Committee opinion no 611: method for estimating due date. Obstet Gynecol. 2014 Oct;124(4):863-866. doi: 10.1097/01.AOG.0000454932.15177.be. PMID 25244460
- [Background] Hanley JA, McNeil BJ. A method of comparing the areas under receiver operating characteristic curves derived from the same cases. Radiology. 1983 Sep;148(3):839-43. doi: 10.1148/radiology.148.3.6878708.
- [Background] Obuchowski NA, McClish DK. Sample size determination for diagnostic accuracy studies involving binormal ROC curve indices. Stat Med. 1997 Jul 15;16(13):1529-42. doi: 10.1002/(sici)1097-0258(19970715)16:133.0.co;2-h. PMID 9249923
- [Background] Buhimschi IA, Christner R, Buhimschi CS. Proteomic biomarker analysis of amniotic fluid for identification of intra-amniotic inflammation. BJOG. 2005 Feb;112(2):173-81. doi: 10.1111/j.1471-0528.2004.00340.x. PMID 15663581
- [Derived] Markenson GR, Saade GR, Laurent LC, Heyborne KD, Coonrod DV, Schoen CN, Baxter JK, Haas DM, Longo S, Grobman WA, Sullivan SA, Major CA, Wheeler SM, Pereira LM, Su EJ, Boggess KA, Hawk AF, Crockett AH, Fox AC, Polpitiya A, Fleischer TC, Critchfield GC, Burchard J, Boniface JJ, Lam GK. Performance of a proteomic preterm delivery predictor in a large independent prospective cohort. Am J Obstet Gynecol MFM. 2020 Aug;2(3):100140. doi: 10.1016/j.ajogmf.2020.100140. Epub 2020 May 17. PMID 33345877